CLINICAL TRIAL: NCT01283958
Title: Study of the Effects of Inhaled Iloprost on Congenital Heart Disease With Eisenmenger Syndrome
Brief Title: The Effects of Inhaled Iloprost on Congenital Heart Disease With Eisenmenger Syndrome
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Song I Yang, Gil Hospital, Gachon University of Medicine
Other Study IDs: no sponsor
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-05

CONDITIONS: Eisenmenger's Syndrome
Keywords: Iloprost, Eisenmenger's syndrome
MeSH Terms: conditions — Eisenmenger Complex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Identification of the pathophysiology associated with Eisenmenger's syndrome has led to the evaluation of targeted therapies. Iloprost, a prostacyclin analogue, is one such targeted therapy used in patients with Eisenmenger's syndrome. The purpose of our study is to assess the effects of inhaled iloprost on patients with Eisenmenger's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients with Eisenmenger's syndrome diagnosed by right side cardiac catheterization

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 12 patients with Eisenmenger's syndrome diagnosed by right side cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-09; Study Completion 2010-05 (Actual)